CLINICAL TRIAL: NCT07046546
Title: Thyroid ARtery Goitre Embolization Trial: A Service Introduction and Safety Assessment
Brief Title: Thyroid Artery Goitre Embolization Trial A Pilot Study Investigating Thyroid Artery Embolisation as a Treatment for Large Thyroid Nodules
Acronym: TArGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Berkshire NHS Foundation Trust (Other Government)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS338447
Record Dates: First submitted 2025-05-02; First posted 2025-07-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Nodule (Benign); Graves Disease; Goitre
Keywords: Thyroid artery embolisation; Benign thyroid nodules
MeSH Terms: conditions — Thyroid Nodule; Graves Disease; Goiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thyroid artery embolization treatment (Experimental): Patient undergoing thyroid artery embolization
  Interventions: Procedure: Thyroid artery embolization

INTERVENTIONS:
Procedure: Thyroid artery embolization — A minimally invasive procedure where one or more thyroid arteries are occluded to shrink the thyroid gland or thyroid nodules
  Other Names: TAE

SUMMARY:
Large non-cancerous thyroid nodules (lumps in the thyroid gland) can cause pressure or discomfort in the neck or cosmetic issues. The standard treatment options include radiofrequency ablation, radioactive iodine, and surgery. Not all patients are suitable however for these treatments, some lumps are too large, or the patients are not fit enough for surgery.

Thyroid artery embolization (TAE) is a new minimally invasive technique (smaller incisions / cuts and shorter recovery time) performed under light sedation. It is used by other European Thyroid Centres, but it hasn't been used in the UK. Embolization means arteries supplying the thyroid gland are blocked by injecting small occlusive particles, like very fine grains of sand that can get stuck in small spaces, preventing blood from passing through. Blocking the thyroid arteries causes the gland to shrink. This provides symptom relief or controls an overactive gland.

We aim to undertake a TAE pilot study to explore the safety of TAE in a UK patient population. We are planning to recruit 10 eligible patients. We will also collect additional data (for example on pain, effectiveness, cost and health related quality of life) to inform a future larger trial comparing TAE to other treatment options.

DETAILED DESCRIPTION:
Justification:

Large thyroid nodules in the neck can cause local pressure symptoms and cosmetic issues. Current treatment options include radioactive iodine (RAI), radiofrequency ablation (RFA) and surgery but larger nodules are difficult to shrink or remove and are associated with risks that some patients find unacceptable such as an underactive thyroid gland which requires life long tablets and surgical scars. Larger nodules are also more difficult to remove surgically.

Thyroid artery embolisation (TAE) is a new procedure for non-cancerous thyroid nodules which are causing local symptoms or hyperthyroidism (overactive thyroid glands). TAE involves blocking thyroid arteries using tiny particles introduced via a small tube (catheter). The tube is guided to the thyroid artery under x-ray guidance. In published studies TAE has been used in small numbers of patients with large thyroid glands where other treatment options are difficult. Evidence shows TAE is safe and improves thyroid function in patients with an overactive gland. TAE also causes gland shrinkage (between 40% to 70%) and improves local neck symptoms (like tightness or pressure), cosmetic appearance and quality of life.

Early research indicates TAE is promising but wider use of the procedure is limited by a lack of high-quality research with larger numbers of patients. It has also never been evaluated in the NHS or UK. We therefore aim to undertake the first UK feasibility study into TAE to primarily evaluate safety. This study will help inform a future larger trial to understand how effective TAE is.

Methodology:

Single site study at Royal Berkshire NHS Foundation Trust.

10 patients will be recruited to the study. Participants will have been diagnosed with an enlarged thyroid gland which is causing local neck symptoms (e.g. pressure or tightness), cosmetic issues or thyroid overactivity.

1. Patient will be first seen and assessed by the ENT team or Interventional Radiology Consultants who confirm the patient has non-cancerous thyroid nodules and requires treatment for their thyroid disease. This is standard care.
2. All patients are then seen by the ENT team (if not already seen). The ENT team consider whether the patient is suitable for study inclusion and discuss possible study participation with the patient. The ENT team provide a study patient information sheet (PIS) and after care advice sheet at this time. With the patients permission the ENT team provides the patients contact details to the research study team (via hospital email or electronic messaging). The ENT team will also document study discussion in the patients electronic records. (10 minutes)
3. Study team contacts the patient by telephone and discusses the study. Patient questions addressed. Telephone consent obtained. Patient sent a copy of the consent form prior to their study pre-assessment clinic (by email or paper form by post). (20 minutes)

   If individuals require more time to consider participation they will be contacted again at an agreed time.
4. Potential participants will attend a screening visit in the Interventional Radiology department at RBFT. The following investigations would then be performed / arranged: ultrasound, needle tests of thyroid gland, CT and blood tests.

(40 minutes).

5. Study team (principle investigator) assesses all results of the screening visit. If the patient meets study inclusion criteria, study team (research nurse) liaises with Radiology booking team and arranges TAE treatment date. Patient and GP informed by letter/email. Patient will be sent a quality of life questionnaire by post or email (30 minutes).

If any results indicate TAE is unsuitable (e.g. abnormal needle test result) the patient will be referred back to the ENT team for standard care.

6. Study intervention (TAE) performed. (3 hours which includes arrival, admission and procedure time).

(Please note an external expert who is highly experienced in TAE will be present for the first two cases. They will only observe and advise where necessary)

9. Patient monitored in Radiology recovery area for 4 hours after procedure (4 hours)

10. Patient admitted to ENT ward for overnight observations and then discharged by research team the following day (approximately 16 to 24 hours)

11. One week post procedure telephone appointment: Analgesia questionnaire and adverse event score completed (can also be sent by post or email and returned by post or email if required). (30 minutes)

12. 3 months post procedure appointment: Quality of life questionnaires; Local symptom and cosmetic scores (out of 10); Thyroid function blood tests; Thyroid volume on ultrasound or CT arranged if required (1h)

13. 6 months post procedure appointment: Quality of life questionnaires; Local symptom and cosmetic scores (out of 10); Thyroid function tests; Thyroid volume on ultrasound or CT arrange if required (1h)

(Please note clinical assessment / evaluations will be undertaken outside these time points if clinically indicated).

ELIGIBILITY:
Inclusion Criteria:

* The participant may enter the study if ALL of the following apply:

  * Adults over 18 years of age willing and able to give informed consent.
  * Symptomatic or cosmetically distressing benign nodular thyroid disease with or without intrathoracic extension and with or without hyperthyroidism. Or auto-immune hyperthyroidism (Graves disease).
  * Single nodular goitre causing local mass effect warranting treatment or multi-nodular goitre
  * TIRADS score 1, 2 and 3 nodules (benign or mildly suspicious) as assessed by ultrasound.
  * FNA confirmed benign disease (x2 FNA Thy2 (benign) result required for TR3 nodules, 1x FNA if nodule classified TR2 or less). FNA performed on most high grade nodule or if equal grade then largest nodule.
  * No enlarged / suspicious neck lymphadenopathy on ultrasound.
  * Patient willing to undergo thyroid nodule embolization in preference to other viable treatment options after discussion with Consultant ENT surgeon and / or Consultant Interventional Radiologist. TAE can also be performed as a bridge to surgery, Radiofrequency ablation or Radioactive iodine. Patients may also be unsuitable or unfit for other treatment options.
  * Patient able to lay on the angiography table flat with one or two pillows, and can lay comfortably with 30 degrees or less of head elevation for a minimum of two hours.

Exclusion Criteria:

* The participant may enter the study if ALL of the following apply:

  * Adults over 18 years of age willing and able to give informed consent.
  * Symptomatic or cosmetically distressing benign nodular thyroid disease with or without intrathoracic extension and with or without hyperthyroidism. Or auto-immune hyperthyroidism (Graves disease).
  * Single nodular goitre causing local mass effect warranting treatment or multi-nodular goitre
  * TIRADS score 1, 2 and 3 nodules (benign or mildly suspicious) as assessed by ultrasound.
  * FNA confirmed benign disease (x2 FNA Thy2 (benign) result required for TR3 nodules, 1x FNA if nodule classified TR2 or less). FNA performed on most high grade nodule or if equal grade then largest nodule.
  * No enlarged / suspicious neck lymphadenopathy on ultrasound.
  * Patient willing to undergo thyroid nodule embolization in preference to other viable treatment options after discussion with Consultant ENT surgeon and / or Consultant Interventional Radiologist. TAE can also be performed as a bridge to surgery, Radiofrequency ablation or Radioactive iodine. Patients may also be unsuitable or unfit for other treatment options.
  * Patient able to lay on the angiography table flat with one or two pillows, and can lay comfortably with 30 degrees or less of head elevation for a minimum of two hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | 18 months
  To undertake thyroid artery embolisation (TAE) pilot study and make a preliminary (non-powered) evaluation of TAE safety.
  The primary end-point is safe treatment with TAE of 10 patients over an 18 month period.

SECONDARY OUTCOMES:
Recruitment | 18 months
  Assess difficulties in recruiting patients by monitoring patient recruitment to time and target
Procedural pain | 1 week
  Procedural pain (Pain score, analgesia use and adverse event recording at 1 week (7 to 10 days).
Procedural outcome | 3 and 6 month follow up
  Pre-TAE and 3 and 6 months post TAE: Procedural effectiveness (patient reported symptom and cosmetic scores, thyroid function blood tests, ultrasound (+/-CT assessment) before and at time intervals after TAE).
  Pre-TAE and 3 and 6 months post TAE: Health related quality of life impact (Questionnaires before and at time intervals after procedure)
Cost | 24 months
  At study end: Assess cost effectiveness - analysis by Trust financial analyst will be undertaken

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Berkshire Hospital, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators aim to disseminate study findings through presentation and publication